CLINICAL TRIAL: NCT03691701
Title: Pilot to Examine Risk and Feasibility of Remote Management of BP From Childhood Into Early Adulthood
Acronym: PERFORMANCE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17-22758
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Chronic Kidney Diseases; Hypertension; Blood Pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Strict SBP Target (Experimental): Home SBP target < 120 mmHg or 90th percentile for age and height (whichever is lower)
  Interventions: Other: strict blood pressure control
- Usual SBP Target (No Intervention): Usual care, no home SBP target

INTERVENTIONS:
Other: strict blood pressure control — Home SBP target < 120 mmHg or 90th percentile for age and height (whichever is lower)
  Arms: Strict SBP Target

SUMMARY:
Hypertension is an increasingly common problem in children, especially among those who are obese or with diabetes and chronic kidney disease. This study is a pilot randomized controlled trial designed to test whether improved blood pressure control can be achieved with the use of remote home blood pressure monitoring in children with uncontrolled blood pressure.

DETAILED DESCRIPTION:
Hypertension is an increasingly common problem in children, especially among those who are obese or with diabetes and chronic kidney disease. This study is a pilot randomized controlled trial designed to test whether improved blood pressure control can be achieved with the use of remote home blood pressure monitoring in children with uncontrolled blood pressure. Study investigators will randomize 60 children who have elevated BP (defined as receipt of ≥1 anti-hypertensive agent or office SBP ≥90th percentile) to either home BP monitoring with a home SBP target of < 90th percentile or less than 120 mm Hg, which ever is lower (intervention group) versus usual care group in 2:1 ratio. This study aims to (1) compare the safety of BP lowering in intervention versus usual care patients, (2) determine the efficacy of the intervention and provide estimates for the refinement of sample size determination for an eventual full-scale trial, and (3) assess the feasibility and acceptability of the intervention, recruitment rates, and barriers to trial completion.

ELIGIBILITY:
Inclusion Criteria:

* must be receiving at least one anti-hypertensive agent or have an office SBP ≥120 mmHg or >90th percentile for age, sex or height at the time of the screening visit
* have a mid-arm circumference between 22-37cm (BP cuff size limitation)
* able to provide consent to participate in our study
* able to use smartphones, or able to use any phone to call or text our study personnel with home BP readings. If participant does not have a smartphone, they will be allowed to call, text, or e-mail home BP readings on a weekly basis instead.

Exclusion Criteria:

We will exclude those who:

* are or are planning to become pregnant, due to inability to take multiple classes of anti-hypertensive agents
* are marginally housed, due to concerns regarding routine follow-up
* are actively participating in a different interventional trial that may affect blood pressure
* are unwilling to consent to participate
* institutionalized individuals or prisoners
* are actively abusing illicit drugs or alcohol
* have a history of poor or doubtful compliance (e.g., frequently missed appointments)
* have office SBP >170 mmHg
* are already taking ≥5 anti-hypertensive medications (any classes, including diuretics)
* have cognitive impairment prohibiting participation in the study

Ages: 13 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Achieved Blood Pressure | Time Frame: Months 4-12

SECONDARY OUTCOMES:
Number of participants screened who enroll in trial | Months 0-12
  Feasibility of enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Ku, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No